CLINICAL TRIAL: NCT04184310
Title: Modified Perineal Linear Stapler Resection for External Rectal Prolapse: a Novel Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, osama khalil, assistant profeosser, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR-170133-1
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- old patient with rectal prolapse (Experimental): old co-morbid patient with complete rectal prolapse unfit for abdominal operation
  Interventions: Other: Modified perineal linear stapler resection for external rectal prolapse

INTERVENTIONS:
Other: Modified perineal linear stapler resection for external rectal prolapse — After anesthesia and patient position, the prolapse was pulled out Two vertical incision were made in both the inner and outer walls of the prolapse (at 3and 9 o'clock)1-2 cm in size approximately 2 cm above the dentate line. We used a reloadable linear cutter stapler (GIA 100mm Covidien, Mansfield, Mass., USA) passing through the tunnel to cut the anterior aspect of the prolapse . Then, after reload the stapler by the new cartridge, we used it to do the same for posterior wall and the prolapsed rectum was completely transected . We ensure that the stapler did not fire at the dentate line to avoid post-operative pain. Multiple 3-0 PDS intermittent full thickness sutures were done for hemostasis. The prolapsed rectum falls back into place spontaneously.

SUMMARY:
from December 2016 to July 2019, 36 elderly co-morbid patients with rectal prolapse were involved in this study which is performed in the GIT surgery unit of Zagazig University Hospital. the investigators used a modified linear stapler resection technique for the rectal prolapse. Postoperative follow up was done for one year to evaluate functional outcome, operative time, hospital stay and complications

DETAILED DESCRIPTION:
The study was done in the GIT Unit of the General Surgery Department of Zagazig University Hospital in the period from December 2016 to July 2019. The hospital Institutional Review Board approved the study protocol. Thirty-six old, co-morbid and short life expectancy patients were included in the sample. They were evaluated for PSP. Informed consent was signed by all patients or first-degree relatives after full discussion of the advantage and disadvantage of the operation. Preoperative bimanual examination was done for rectal prolapse to rule out enterocele or cystocele and this was confirmed by MRI. The routine preoperative evaluation was done for all patients (physical examination, complete blood tests, ECG and chest x-ray). Bowel preparation was done for all patients.

Regarding bowel function, all patients were evaluated for fecal incontinence by Wexner score and for constipation by Rome II criteria. Prophylactic intravenous cephalosporin and metronidazole was given one hour before operation. The operation was done under spinal anesthesia in the lithotomy position with slight Trendeleburg to prevent trapping of abdominal organs between walls of rectum. All operations were done by the same surgical members of the unit. Hospital stay, Intraoperative and postoperative complications were recorded. All patients started oral fluids in the second day. Follow up was done for patients every 1,3,6,9 and 12 months in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* old age
* complete rectal prolapse
* co-morbid ASA I to III

Exclusion Criteria:

-

Ages: 48 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
treatment of rectal prolapse | 30 dyas
  patients satisfaction after operation - no mass coming form anus - no previous complications like bleeding and constipation

SECONDARY OUTCOMES:
post operative complications | one year
  bleeding - infection - constipation-incontinence- recurrence

CONTACTS AND LOCATIONS:
Overall Officials: osama khalil, Ph.d, Principal Investigator — assistant professor
Locations (1):
- Zagazig Unversity, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided